CLINICAL TRIAL: NCT02535494
Title: Risks and Benefits of Overdose Education and Naloxone Prescribing to Heroin Users
Brief Title: Risks and Benefits of Naloxone Prescribing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Indivior Inc. (Industry); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Jermaine Jones, Assistant Professor of Clinical Neurobiology, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 6723; R01DA035207 (NIH)
Record Dates: First submitted 2015-08-25; First posted 2015-08-28 (Estimated); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Opioid Overdose
MeSH Terms: conditions — Opiate Overdose

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard Training (No Intervention): Participants receive our standard overdose training.
- Extensive Training (Experimental): Participant receives an more in-depth, extensive training concerning opioid overdose.
  Interventions: Other: Extensive training
- Extensive Training w/ Significant Other (Experimental): Participant and their significant other both receive a more in-depth, extensive training concerning opioid overdose.
  Interventions: Other: Extensive training

INTERVENTIONS:
Other: Extensive training — We have developed a more in-depth education package to help participants better recognize and respond to an opioid overdose.
  Arms: Extensive Training; Extensive Training w/ Significant Other

SUMMARY:
This investigation is one of the first large-scale, prospective attempts to obtain data on the effectiveness of naloxone distribution among opioid-abusing populations at high risk of unintentional opioid poisoning. Specifically, opioid abusers will be recruited from drug detoxification sites as well as those accessing services at needle exchange programs. All participants (N=700) will receive the standard opioid overdose education and naloxone. One third of the participants will be randomized to receive additional in-depth psychosocial education focusing on recognition and prevention of opioid overdose, and appropriate use of naloxone. Another third of the participants will receive the extensive training and be required to engage a spouse, partner, relative, or friend in this supplementary intervention. The investigators plan to randomize individuals to each group [Treatment as Usual (TAU) vs. Extensively Trained (ET) vs. Extensively Trained with a Significant Other (ETwSO)] and, through continued follow up over one year, the investigators will compare self-reported overdose reversal attempts (with and without naloxone use), naloxone-related adverse events, and changes in patterns of heroin and other drug use.

DETAILED DESCRIPTION:
Study Design A significant cause of mortality among opioid users is overdose, which commonly occurs following voluntary (opioid detoxification) or involuntary (incarceration) opioid abstinence. For the purposes of the current application, opioid overdose is defined as use of an opioid in an amount that results in over-sedation and/or respiratory depression requiring intervention by medical or non-medical persons. Nearly 85% of overdoses occur in the presence of a witness. Common methods of intervention by individuals without medical training are ineffective techniques such as shaking the victim or injecting salt water. Naloxone is an opioid antagonist that has long been used successfully by trained medical personnel during emergency resuscitation following opioid overdose. In an effort to reduce fatal and non-fatal opioid overdose, a number of states are implementing programs in which non-medical personnel are provided brief instruction in recognizing the signs of opioid overdose and administering naloxone. However, most of the existing programs are not designed to collect empirical data on the safety and effectiveness of this intervention. Reporting of naloxone use is voluntary and without incentive, and the experience of those who have been trained and prescribed naloxone is not followed.

The proposed investigation will be one of the first large-scale, prospective attempts to obtain data on the effectiveness of naloxone distribution among opioid-abusing populations at high risk of unintentional opioid poisoning. Specifically, opioid abusers will be recruited from drug detoxification sites as well as those accessing services at needle exchange programs. All participants (N=700) will receive the standard opioid overdose education and naloxone. One third of the participants will be randomized to receive additional in-depth psychosocial education focusing on recognition and prevention of opioid overdose, and appropriate use of naloxone. Another third of the participants will receive the extensive training and be required to engage a spouse, partner, relative, or friend in this supplementary intervention. We plan to randomize individuals to each group [Treatment as Usual (TAU) vs. Extensively Trained (ET) vs. Extensively Trained with a Significant Other (ETwSO)] and, through continued follow up over one year, we will compare self-reported overdose reversal attempts (with and without naloxone use), naloxone-related adverse events, and changes in patterns of heroin and other drug use. In addition to comparing outcome variables in the TAU, ET and ETwSO groups prospectively, we will analyze data collected before study initiation to compare fatal and non-fatal opioid overdose rates in neighborhoods with facilities that offer overdose prevention training and naloxone to those that do not, using data provided by our collaborators at the New York City (NYC) Department of Health and Mental Hygiene (DOHMH).

Specific Aims and Hypotheses

* Primary Aim (Prospective Study): Determine the extent to which additional psychosocial intervention can improve the effectiveness of current overdose prevention training as measured by:
* increased frequency of naloxone use (ETwSO > ET > TAU)
* decreased number of opioid overdoses (ETwSO < ET < TAU)
* improved recognition of opioid overdose and naloxone indication knowledge (increased BORRA scores; ETwSO > ET > TAU)
* Secondary Aim (Prospective Study): Determine the potential harms of this novel naloxone-prescribing practice as measured by:
* proportion of participants calling 911 in response to an overdose, compared to participants' recent history of calling 911 in response to an overdose
* risky drug use behavior (e.g. increased heroin/prescription opioid use, increased use of illicit drug combinations) following training, compared to pre-training

Outcome Measures

Primary Outcome Measures (Prospective Study): Determine the extent to which additional psychosocial intervention can improve upon the effectiveness of current overdose prevention training by: 1) increasing the frequency of naloxone use among ET participants (continuous variable); 2) decreasing the number of lethal opioid overdoses witnessed and experienced by the ET group (continuous variable); 3) improving accurate recognition of opioid overdose and naloxone indication knowledge (increased Brief Overdose Recognition and Response Assessment (BORRA) score among ET participants (continuous variable). These variables will be assessed repeatedly over the course of 1 year at: baseline (BL), immediately post-training (T0), 1-, 3-, 6- and 12-months (T1, T3, T6, and T12). The frequency of naloxone use and outcomes of the overdose reversal attempts will be measured at T1, T3, T6, and T12 only.

Secondary Outcome Measures (Prospective Study): Evaluate the potential harms of this novel naloxone-prescribing practice as assessed by: 1) decreased proportion of 911 calls in response to an overdose, compared to participants' previous history of calling 911 while witnessing an overdose (continuous variable); 2) changes in the use of illicit opioids, other illegal drugs, or drug combinations following training (longitudinal continuous variable); 3) prevalence of adverse events related to naloxone administration by non-medical personnel (continuous variable).

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 21 to 65 years
* Has met DSM-V criteria for moderate-severe opioid use disorder within the past 6-months, actively using heroin, prescription opioids, or has detoxified within the last 3 months.
* In otherwise good health based on medical history and laboratory tests
* Able to provide informed consent and comply with study procedures
* Able to fluently speak and read English
* Able to identify a spouse, friend or relative who willing to serve as their "significant other"

Exclusion Criteria:

* Active psychiatric disorder that might interfere with participation or make participation hazardous, including DSM-V organic mental disorder, psychotic disorder, or bipolar disorder with mania
* Previous Basic Cardiac Life Support or First-Aid training
* Active treatment with extended-release naltrexone (Vivitrol) for alcohol or opioid dependence
* Naloxone training for opioid overdose prevention in the previous 2 years (Clinical Interview)

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 405 (Actual)
Dates: Start 2014-07; Primary Completion 2021-05 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Likelihood of Naloxone Use | 1 year
  Determine the extent to which additional psychosocial intervention can improve upon the effectiveness of current overdose prevention training by increasing the frequency of naloxone use
Overdose Reversal Outcome | 1 year
  Determine the extent to which additional psychosocial intervention can improve the ability of the training to decrease the number of lethal opioid overdoses.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra D Comer, PhD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jones JD, Campbell AN, Brandt L, Metz VE, Martinez S, Wall M, Corbeil T, Andrews H, Castillo F, Neale J, Strang J, Ross S, Comer SD. A randomized clinical trial of the effects of brief versus extended opioid overdose education on naloxone utilization outcomes by individuals with opioid use disorder. Drug Alcohol Depend. 2022 Aug 1;237:109505. doi: 10.1016/j.drugalcdep.2022.109505. Epub 2022 May 23. PMID 35709575